CLINICAL TRIAL: NCT03439787
Title: The Effect of the Popliteal Plexus Block on Postoperative Pain After Total Knee Arthroplasty - a Randomized, Controlled, Double-blinded Study
Brief Title: Popliteal Plexus Block for Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Methodological problems/problems in the study design (competing pain and a placebo effect). No serious adverse events or other safety issues
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol_PPB_TKA_31122017; 2017-005180-40 (EudraCT Number)
Record Dates: First submitted 2018-01-18; First posted 2018-02-20 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
Keywords: Arthroplasty, Replacement, Knee; Anesthetics, Local; Pain, Postoperative; Nerve Block; Bupivacaine; Epinephrine
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Popliteal Plexus Block (Active Comparator): 10 ml Bupivacaine-Epinephrine 0.5%-1:200,000 Injectable Solution
  Interventions: Drug: Bupivacaine-EPINEPHrine 0.5%-1:200,000 Injectable Solution
- Placebo Popliteal Plexus Block (Placebo Comparator): 10 ml Sodium Chloride 0.9 %
  Interventions: Other: Sodium Chloride 0.9 %

INTERVENTIONS:
Drug: Bupivacaine-EPINEPHrine 0.5%-1:200,000 Injectable Solution — 10 ml
  Other Names: Marcain-adrenaline
  Arms: Active Popliteal Plexus Block
Other: Sodium Chloride 0.9 % — 10 ml
  Arms: Placebo Popliteal Plexus Block

SUMMARY:
This study aims to assess the analgesic effect of the popliteal plexus block as a supplement to a femoral triangle block in patients undergoing total knee arthroplasty

DETAILED DESCRIPTION:
A femoral triangle block (FTB) effectively anesthetizes the anterior group of nerves innervating the knee (infrapatellar branch of the saphenous nerve, the medial femoral cutaneous nerve and the terminal branch of the medial vastus muscle nerve). However, the posterior group of nerves innervating the knee joint is not covered with an FTB, and therefore most patients complain of significant, opioid-requiring pain despite a successful FTB.

The posterior group consists of the popliteal plexus, which is derived from the tibial nerve and the posterior branch of the obturator nerve. The popliteal plexus is located in the popliteal fossa, where it entwines the popliteal artery and vein. Recent cadaver studies have suggested that an injection into the distal part of the adductor canal will spread to the popliteal fossa (PubMed Identifier (ID): 28937534; PubMed ID: 27442773).

This study aims to assess the analgesic effect of the popliteal plexus block (PPB) as a supplement to a femoral triangle block (FTB) after total knee arthroplasty (TKA).

In the study all patients will receive an FTB with 10 ml bupivacaine-epinephrine (0.5%-1:200,000) with the addition of 0.5 ml Dexamethasone (4 mg/ml).

All patients are postoperatively observed for the development of significant pain (NRS > 3) in the primary observation period (POP) defined as: a 3-hour observation period starting at the return of completely normal cutaneous sensation (lateral thigh and lateral side of the lower leg) after spinal anesthesia. If the patient reports pain (NRS > 3) in the POP, the patient will be randomized to the study treatment - a PPB with 10 ml bupivacaine-epinephrine or 10 ml saline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 50 years of age at screening
* Scheduled to undergo primary total knee arthroplasty in spinal anesthesia
* Normal sensory function at the lateral part of the thigh and lower leg
* American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
* Able to provide informed consent

Exclusion Criteria:

* Unable to cooperate and follow the study protocol
* Communication problems
* Allergic towards any medical product administered in the study
* Diabetes requiring medical treatment
* Pregnancy (a pregnancy test will be conducted on all women of childbearing potential prior to inclusion in the study. A positive test result will result in exclusion from the study)
* Preoperative opioid treatment (dosed > once daily)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Success of the popliteal plexus block (PPB) | 60 minutes after placement of the PPB
  Success of the PPB is defined as the proportion of patients with significant postoperative pain (NRS > 3) after FTB, who drop in pain score to NRS ≤ 3 after PPB and maintain NRS ≤ 3 without any opioids until 60 minutes after PPB

SECONDARY OUTCOMES:
Onset time of the PPB | The pain scores after PPB are evaluated every 5 minutes until 15 minutes after PPB and hereafter every 15 minutes until 60 minutes after PPB
  The onset time is defined as the time from withdrawal of the block needle and until the patient reports NRS ≤ 3. The maximal onset time is defined as 60 minutes
The effect of the PPB on cutaneous sensation | Baseline and 2 hours after the placement of the PPB
  Performed as a pinprick test on the lateral aspect of the lower leg. Sensation to pinprick is graded on a 3-point scale: 0 = no sensation, 1 = reduced sensation and 2 = normal sensation to pinprick compared to the contralateral side
The effect of PPB on isometric muscle strength of the he dorso- and plantar flexors of the ankle joint | Baseline and 2 hours after the placement of the PPB
  Dorsal and plantar flexion of the foot is measured as the maximum voluntary isometric contraction (MVIC). During the test, a handheld dynamometer is kept immobile and the patient is asked to push against the dynamometer with maximal force and maintain this maximal pressure for 5 seconds. The MVIC is measured three times, separated by a 30-second pause, and the highest of the three MVIC values is registered
Opioid consumption from 0-4 hours | Subjects receiving PPB: From after PPB placement and up until 4 hours after PPB. Subjects not receiving PPB: From the end of the primary observation period (POP) and up until 4 hours after the end of the POP
  Registered from the electronic patient record
Opioid consumption from 4-24 hours | Subjects receiving PPB: From 4 hours after PPB placement and up until 24 hours after PPB. Subjects not receiving PPB: From 4 hours after the end of the POP and up until 24 hours after the end of the POP
  Registered from the electronic patient record
Pain scores (Numerical Rating Scale, NRS, 0-10 where 0 is "no pain" and 10 is "worst pain imaginable" | For subjects receiving a PPB, pain scores will be performed 2, 4 and 24 hours after PPB. For subjects not receiving a PPB, final pain scores will be made at the 24 hrs follow-up visit
  The patient is asked about the worst pain since last test time
Pain localization | Subjects with NRS > 3: when significant pain is reported during the POP; 15 and 60 min after PPB; at any increase in NRS score at any time during the 60 min after PPB; 2, 4 and 24 hrs after PPB. For subjects with NRS ≤ 3: at the 24 hrs follow-up visit
  Evaluated using a systematic questionnaire
The number of patients requiring a PPB | All patients receive an FTB and are observed postoperatively for the development of NRS > 3 during the primary observation period (POP) defined as: A 3-hour observation period starting at the return of normal cutaneous sensation after spinal anesthesia
  The number of patients experiencing NRS > 3 as a proportion of all patients with femoral triangle block (FTB)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte R Sørensen, MD, Principal Investigator — Silkeborg Regional Hospital
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. The Optimal Analgesic Block for Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):711-719. doi: 10.1097/AAP.0000000000000485. PMID 27685346
- [Background] Wong WY, Bjorn S, Strid JM, Borglum J, Bendtsen TF. Defining the Location of the Adductor Canal Using Ultrasound. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):241-245. doi: 10.1097/AAP.0000000000000539. PMID 28002228
- [Background] GARDNER E. The innervation of the knee joint. Anat Rec. 1948 May;101(1):109-30. doi: 10.1002/ar.1091010111. No abstract available. PMID 18915634
- [Background] Abdallah FW, Chan VW, Gandhi R, Koshkin A, Abbas S, Brull R. The analgesic effects of proximal, distal, or no sciatic nerve block on posterior knee pain after total knee arthroplasty: a double-blind placebo-controlled randomized trial. Anesthesiology. 2014 Dec;121(6):1302-10. doi: 10.1097/ALN.0000000000000406. PMID 25099748
- [Background] Abdallah FW, Madjdpour C, Brull R. Is sciatic nerve block advantageous when combined with femoral nerve block for postoperative analgesia following total knee arthroplasty? a meta-analysis. Can J Anaesth. 2016 May;63(5):552-68. doi: 10.1007/s12630-016-0613-2. Epub 2016 Feb 19. PMID 26896282
- [Background] Runge C, Borglum J, Jensen JM, Kobborg T, Pedersen A, Sandberg J, Mikkelsen LR, Vase M, Bendtsen TF. The Analgesic Effect of Obturator Nerve Block Added to a Femoral Triangle Block After Total Knee Arthroplasty: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):445-51. doi: 10.1097/AAP.0000000000000406. PMID 27171822
- [Background] McNamee DA, Parks L, Milligan KR. Post-operative analgesia following total knee replacement: an evaluation of the addition of an obturator nerve block to combined femoral and sciatic nerve block. Acta Anaesthesiol Scand. 2002 Jan;46(1):95-9. doi: 10.1034/j.1399-6576.2002.460117.x. PMID 11903080
- [Background] Taha AM. Brief reports: ultrasound-guided obturator nerve block: a proximal interfascial technique. Anesth Analg. 2012 Jan;114(1):236-9. doi: 10.1213/ANE.0b013e318237fb40. Epub 2011 Oct 24. PMID 22025494
- [Background] Goffin P, Lecoq JP, Ninane V, Brichant JF, Sala-Blanch X, Gautier PE, Bonnet P, Carlier A, Hadzic A. Interfascial Spread of Injectate After Adductor Canal Injection in Fresh Human Cadavers. Anesth Analg. 2016 Aug;123(2):501-3. doi: 10.1213/ANE.0000000000001441. PMID 27442773
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Runge C, Moriggl B, Borglum J, Bendtsen TF. The Spread of Ultrasound-Guided Injectate From the Adductor Canal to the Genicular Branch of the Posterior Obturator Nerve and the Popliteal Plexus: A Cadaveric Study. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):725-730. doi: 10.1097/AAP.0000000000000675. PMID 28937534
- See also: The pilot study on which the current study is based — https://clinicaltrials.gov/ct2/show/NCT03198403?term=NCT03198403&rank=1